CLINICAL TRIAL: NCT03787641
Title: Sysytematic Evaluation of Heparin and Protamine in Cardiac Surgery
Brief Title: Systematic Evaluation of Protamine Doze in Cardiac Surgery
Acronym: HART
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Ravi Taneja, Associate Scientist, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 107681
Record Dates: First submitted 2016-05-13; First posted 2018-12-26 (Actual); Last update posted 2018-12-31 (Actual); Status verified 2018-12

CONDITIONS: Cardiac Surgery With Cardiopulmonary Bypass
Keywords: cardiopulmonary bypass; heparin; protamine; anti-IIa assay; anti-Xa assay; activated clotting time
MeSH Terms: interventions — Protamines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Protamine doze (Other): Protamine Sulfate will be administered through an infusion pump in aliquots at a predefined rate (25 mg/min). Blood samples will be withdrawn after each aliquot and quantified for anti-Xa, IIa and ACT.
  Interventions: Drug: Protamine Sulfate

INTERVENTIONS:
Drug: Protamine Sulfate — Protamine Sulfate will be administered via an infusion pump to administer a 50 mg test doze, then 100 mg after 5 min waiting period. Following blood samples, additional alliquots of 50 mg will be measured to a maximum of 300 mg.

SUMMARY:
The precise amount of protamine required to neutralize unfractionated heparin (UFH) remains unknown. This study will systematically identify the doze needed to neutralize UFH following cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
The precise dose of protamine needed to neutralize unfractionated heparin (UFH) is unknown. Research suggests that low dose protamine is associated with decreased need for transfusions in cardiac surgery. The ATS guidelines recommend that half of the total UFH dose given for cardiopulmonary bypass (CPB) should be neutralized with protamine. However, it is unknown if this is routinely followed by anesthesiologists. Furthermore, the reference standard for UFH has changed recently and it is unknown how this has affected the dose of protamine in the perioperative period. Protamine does have a very short life and heparin rebound occurs very commonly.

It is common practice to divert the suctioned mediastinal blood following CPB while the patient is still anticoagulated. The traditional practice is that once half dose protamine has been given, suction to the cardiotomy reservoir is turned off. All surgical field blood loss is then diverted to wall suction. The inherent risk of letting too much protamine into the CPB reservoir is that UFH therein may get neutralized and predispose to clot formation in the venous reservoir. This precludes an emergency 'crash' on to CPB, should that be required for some reason. Experience of the Investigators indicates that most surgeons will turn off suction leading to the cardiotomy reservoir once half the total protamine dose has been administered. The concern with this is that "half dose" protamine may be quite different for different anesthesiologists.

The research investigators hypothesize low dose protamine is sufficient to neutralize the effects of UFH as monitored through activated clotting time (ACT). Anesthesiologists administer varying doses of protamine to neutralize UFH in cardiac surgery and the rationale behind such decisions is unclear.

Thus, the primary objective of this study is to evaluate the dose of protamine required to neutralize UFH following CPB. Secondary objectives are 1) to assess the amount of protamine needed to neutralize UFH in intravenously administered cardiotomy reservoir blood. 2) To examine the amount of residual heparin postoperatively in the cardiac surgery ICU; 3) to examine, through semi-structured interviews, the decision-making processes involved in managing (anti)coagulation in cardiac surgery.

ELIGIBILITY:
Inclusion Criteria:

* Elective cardiac surgery patients > 18 years age who can provide written consent for the study.

Exclusion Criteria:

* History of any known coagulopathies, liver dysfunction, previous cardiac surgery, preoperative abnormal coagulation profiles, recent exposure to heparin (unfractionated or low molecular weight), warfarin, clopidogrel or other direct thrombin inhibitors in the preceding 7 days.
* History of heparin resistance
* History of adverse reactions to protamine
* Patients identified as having heparin resistance
* Anticipated CPB time > 2-2.5 hrs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in heparin activity | Duriing surgery (at baseline, before and after protamine adminitration following cardiopulmonary bypass). Samples will also be quantified at Intensive Care Unit (ICU) admission and 4 hours following ICU admission.
  The functional activity is ideally measured via its ability to accelerate the inhibition of activated coagulation enzymes IIa (thrombin) and Xa respectively.
  These tests are available commercially as ELISA kits. Briefly, an excess of coagulation factor IIa or Xa respectively is added to the sample and residual anti-IIa/Xa activity is quantified with a synthetic chromogenic substrate.
Change in Activated Clotting time (ACT) | Duriing surgery (at baseline, before and after protamine adminitration following cardiopulmonary bypass).
  ACT is the standard point of care test used in cardiac surgery. Blood is added to a tube containing predefined amount of coagulation accelerator (available commercially) and heparin activity is measured by prolongation or neutralization of ACT

SECONDARY OUTCOMES:
Rationale for choosing a certain doze of protamine | During surgery. (Average cardiac surgery lasts for 4-6 hours)
  Anesthesiologists will undergo semi-structured face to face interviews and asked their rationale for choosing a certain doze of protamine

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Derived] Taneja R, Szoke DJ, Hynes Z, Jones PM. Minimum protamine dose required to neutralize heparin in cardiac surgery: a single-centre, prospective, observational cohort study. Can J Anaesth. 2023 Feb;70(2):219-227. doi: 10.1007/s12630-022-02364-4. Epub 2022 Dec 5. PMID 36471142